CLINICAL TRIAL: NCT00730587
Title: Development of a Body Composition Method for Infants and Children
Brief Title: Study of Body Composition Methodology in Young Children (InfantPod)
Status: Withdrawn | Type: Observational
Why Stopped: This study will not be conducted. A new study is replacing this one.
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); University of Arkansas (Other)
Responsible Party: Aline Andres, Ph.D., Universtiy of Arkansas for Medical Science
Other Study IDs: 105169
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Nutrition; Body Fat; Infant; Healthy Babies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine will be collected from all study participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Full-term healthy infants ages 5 months to 3 years.

SUMMARY:
The InfantPod study is a cross-sectional study designed to determine how practical and precise a body composition method is for measuring body fat and lean tissue in infants and children ages 5 months to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children between ages of 5 months and 3 years

Exclusion Criteria:

* Child that has any condition that may affect growth
* Child that has any chronic disease
* Child that has any carbohydrate metabolism disorder
* Child that takes any medications that may interfere with study parameters as determined by the investigator

Ages: 5 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children in the greater Little Rock area.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States